CLINICAL TRIAL: NCT01340079
Title: Virtual World Health Behavior Counseling for Patients With Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1RC1LM010412-01 (NIH)
Record Dates: First submitted 2011-03-16; First posted 2011-04-22 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes mellitus, non-insulin dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual world (Experimental): Virtual world delivery method
  Interventions: Behavioral: virtual world
- face to face (Active Comparator): face to face method of health education
  Interventions: Behavioral: face to face

INTERVENTIONS:
Behavioral: virtual world — health education using virtual world Second Life
  Arms: Virtual world
Behavioral: face to face — health education delivered in face to face groups
  Arms: face to face

SUMMARY:
Comparison of 2 methods of delivery health education for African-American women with Type 2 Diabetes. The two methods are: face to face education in small groups, as compared to delivering the same curriculum in the virtual world, Second Life.

DETAILED DESCRIPTION:
This study will provide health education to African-American women with type 2 diabetes either face to face, or using the Internet. The study seeks to determine how feasible the internet method is for this type of health education, and how it compares to the face to face method. Patients will be recruited from Boston Medical Center. They will do baseline surveys and have blood drawn. They will then be randomized into receiving their diabetes education in a face to face group at BMC, or receiving it online while at home. The online group will receive a computer to access the Internet program and Internet access. Both groups will participate in 8 diabetes education groups, and 4 individual counseling sessions. Subjects will complete surveys before and after the study to measure changes in physical activity, diet, and use of medications, and will have blood tests drawn at BMC before and after the study to measure changes in diabetes control, cholesterol. They will also have blood pressure measured before and after the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with T2DM
2. HbA1c level >= 8.0
3. Currently treated with diet, oral hypoglycemics or insulin. If currently on insulin, must have a history of prior therapy with diet alone or oral hypoglycemic agents
4. African-American origin
5. >= 18 years old
6. Telephone in home or easy access to one
7. Able to understand and participate in the study protocol
8. Functionally capable of meeting the activity goals
9. Understands and can provide informed consent
10. Physician approval to participate in the study.

Exclusion Criteria:

1. History of diabetic ketoacidosis
2. Gestational diabetes
3. Unable or unwilling to provide informed consent
4. Plans to move out of the area within the 12-month study period
5. Required intermittent glucocorticoid therapy within the past 3 months
6. Experienced an acute coronary event (myocardial infarction or unstable angina) within the previous 6 months
7. Has a medical condition that precludes adherence to study dietary recommendations (e.g., Crohn's disease, ulcerative colitis, end-stage renal disease)
8. Has a medical or psychiatric illness (i.e., dementia, psychiatric hospitalization or suicidality within past 5 years or takes an neuroleptic medication). We will not exclude based on history of depression or anxiety or taking anti-depressants or anti-anxiety medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in hemoglobin a1c at 8 weeks after completion of the intervention. | Baseline and 8 weeks after completion of the intervention

SECONDARY OUTCOMES:
Change from Baseline in dietary patterns at 8 weeks after completion of the intervention. | Baseline and 8 weeks after completion of the intervention
Change from Baseline in physical activity at 8 weeks after completion of the intervention. | Baseline and 8 weeks after completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: John M. Wiecha, MD, MPH, Principal Investigator — Boston Medical Center/Boston University Medical Campus; Milagros Rosal, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Rosal MC, Heyden R, Mejilla R, Capelson R, Chalmers KA, Rizzo DePaoli M, Veerappa C, Wiecha JM. A Virtual World Versus Face-to-Face Intervention Format to Promote Diabetes Self-Management Among African American Women: A Pilot Randomized Clinical Trial. JMIR Res Protoc. 2014 Oct 24;3(4):e54. doi: 10.2196/resprot.3412. PMID 25344620